CLINICAL TRIAL: NCT06045234
Title: Temporal Variation of the Exposure to Pesticides in the Employees of the Limoges University Hospital
Acronym: VESTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RI23_0014 (VESTAL)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Toxicology
Keywords: Pesticides; general population; measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pesticide measurement (Experimental)
  Interventions: Other: Urine sampling

INTERVENTIONS:
Other: Urine sampling — Among the 300 people recruited:
  * 300 will each provide 3 urine samples collected on 3 different days during a week (e.g. Monday, Wednesday and Friday)
  * 50 will each provide 3 urine samples collected at sunrise, in the middle and then at the end of the day over a period of 24 hours, on 3 different days during a week (e.g. Monday, Wednesday and Friday).

SUMMARY:
In a sample of 300 employees of the Limoges University Hospital, it is proposed to explore the intraindividual and interindividual variability of urinary concentrations of glyphosate and 320 other pesticides. The employees will fill a questionary in which will allow to explore the relationships between the concentrations, lifestyle and dietary habits.

DETAILED DESCRIPTION:
The general population is exposed to pesticides through the ingestion of food and water. The presence of pesticides in human urine has been demonstrated in numerous studies. Conventionally, biological monitoring studies use an undifferentiated urine sample or the first morning urine. The reliability of measuring a single-point urinary concentration to represent the profile of pesticide exposure in individuals over time is, however, questionable. Rare studies reporting intra-individual outcomes of pesticide exposure have been conducted in specific populations, such as children and pregnant women.

It is proposed to carry out a descriptive biomonitoring study of the urinary concentration of approximately 320 pesticides in a sample of the general population. Among these, the study will focus on glyphosate.

The originality of our study is:

* (i) Exploration of exposure to the main pesticides in a sample of 300 people by measuring urinary concentration by specific and sensitive methods of LC-MS/MS and GC-MS/MS; These 300 subjects will be hospital staff of the Limoges University Hospital.
* (ii) Exploration of the intra-individual variability of exposure by repeating measurements in urine samples taken over a 24-hour period and/or several times over the course of a week;
* (iii) Determination of the frequency of subjects who have potentially been exposed to doses higher than the acceptable daily intake (in particular for glyphosate) (iv) The association of these exposure values with data from a self-administered questionnaire in order to identify the determinants of this exposure
* (V) Estimating the predictability/reliability of a single urine sample to represent this exposure of individuals/populations over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and over.
* Employed by the University Hospital of Limoges.
* Having consented to participate in the study after being informed.

Exclusion Criteria:

- Adult with a professional activity during which he is required to handle or come into contact with glyphosate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
glyphosate overconsumption | 1 week
  Proportion of individuals with an estimated daily consumption of glyphosate greater than the acceptable daily intake of glyphosate

SECONDARY OUTCOMES:
Identification of determinant of exposure to glyphosate | 1 week
  Proportion of individuals with a daily consumption of glyphosate greater than the acceptable daily intake according to socio-demographic determinants(age, sex, profession and socio-professional category)
Identification of determinant of exposure to glyphosate | 1 week
  Proportion of individuals with a daily consumption of glyphosate greater than the acceptable daily intake according to lifestyles (city center, peri-urban, rural )
Identification of determinant of exposure to glyphosate | 1 week
  Proportion of individuals with a daily consumption of glyphosate greater than the acceptable daily intake according to proximity to agricultural activities
Identification of determinant of exposure to glyphosate | 1 week
  Proportion of individuals with a daily consumption of glyphosate greater than the acceptable daily intake according to use of glyphosate at home
Identification of determinant of exposure to glyphosate | 1 week
  Proportion of individuals with a daily consumption of glyphosate greater than the acceptable daily intake according to dietary habits
Coefficient of variation of the glyphosate concentrations | 1 week
  Calculation of the coefficient of variation of the glyphosate concentrations measured 3 times over a period of 24 hours
Intra-individual variability of urinary glyphosate concentrations | 1 week
  Comparison of the average GLP concentrations measured on 3 occasions (at sunrise, in the middle then at the end of the day) over a period of 24 hours.
Impact of urine sample collection schedule on glyphosate concentration measurement | 1 week
  According to the methodology proposed by Wang et al. : a linear mixed-effects model to determine which measure produces the best estimate of exposure; itself obtained by calculating the mean of the observed values.
Identification of determinants of exposure to a panel of around 320 pesticides | 1 week
  Proportion of subjects with a detectable concentration among the 320 pesticides measured by specific LC-MS and GC-MS methods and prevalence of individuals with a detectable concentration according to socio-demographic determinants
Identification of determinants of exposure to a panel of around 320 pesticides | 1 week
  Proportion of subjects with a detectable concentration among the 320 pesticides measured by specific LC-MS and GC-MS methods and prevalence of individuals with a detectable concentration according to lifestyles
Identification of determinants of exposure to a panel of around 320 pesticides | 1 week
  Proportion of subjects with a detectable concentration among the 320 pesticides measured by specific LC-MS and GC-MS methods and prevalence of individuals with a detectable concentration according to proximity to agricultural activities
Identification of determinants of exposure to a panel of around 320 pesticides | 1 week
  Proportion of subjects with a detectable concentration among the 320 pesticides measured by specific LC-MS and GC-MS methods and prevalence of individuals with a detectable concentration according to use of glyphosate at home
Identification of determinants of exposure to a panel of around 320 pesticides | 1 week
  Proportion of subjects with a detectable concentration among the 320 pesticides measured by specific LC-MS and GC-MS methods and prevalence of individuals with a detectable concentration according to dietary habits
Intra-individual variability of urinary 320 pesticides concentrations | 1 week
  Calculation of the coefficient of variation of the concentrations of each of the pesticides (expressed in µg/L or µg/g of creatinine) measured 3 times (at sunrise, in the middle and then at the end of the day) over a period of 24 hours
Impact of urine sample collection schedule on 320 pesticides concentration measurement | 1 week
  Comparison of the average concentrations of each of the pesticides measured on 3 occasions (at sunrise, in the middle and then at the end of the day) over a period of 24 hours. According to the methodology proposed by Wang et al.: a linear mixed-effects model to determine which measure produces the best estimate of exposure; itself obtained by calculating the mean of the observed values.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No